CLINICAL TRIAL: NCT05197712
Title: A Phase 1, Open-label Study to Evaluate the Safety, Tolerability, and Reactogenicity of the Baiya SARS-CoV-2 Vax 2 Vaccine in Healthy Adults
Brief Title: Evaluation of the Safety, Tolerability, and Reactogenicity of the Baiya SARS-CoV-2 Vax 2 Vaccine for COVID-19 Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Baiya Phytopharm Co., Ltd. (Industry)
Collaborators: National Vaccine Institute, Thailand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: Baiya-Vax2-P1
Record Dates: First submitted 2022-01-15; First posted 2022-01-19 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-01

CONDITIONS: COVID-19 Vaccine
Keywords: SARS-CoV-2; SARS-CoV-2 vaccine; COVID-19; COVID-19 Vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 25 μg Baiya SARS-CoV-2 Vax 2 (Experimental): Experimental: 25 μg Baiya SARS-CoV-2 Vax 2, Adult Participants 2 doses of Baiya SARS-CoV-2 Vax 2 (25 μg), each on Day 1 and Day 22 for adult participants (18 - 64 years old)
  Interventions: Biological: 25 Baiya SARS-CoV-2 Vax 2
- 50 μg Baiya SARS-CoV-2 Vax 2 (Experimental): Experimental: 50 μg Baiya SARS-CoV-2 Vax 2, Adult Participants 2 doses of Baiya SARS-CoV-2 Vax 2 (50 μg), each on Day 1 and Day 22 for adult participants (18 - 64 years old)
  Interventions: Biological: 50 Baiya SARS-CoV-2 Vax 2

INTERVENTIONS:
Biological: 25 Baiya SARS-CoV-2 Vax 2 — Intramuscular injection in the deltoid region of 0.5 mL/dose of Baiya SARS-CoV-2 Vax 2 (recombinant SARS-CoV-2 receptor-binding domain fused with FC region of human IgG1 vaccine)
  Arms: 25 μg Baiya SARS-CoV-2 Vax 2
Biological: 50 Baiya SARS-CoV-2 Vax 2 — Intramuscular injection in the deltoid region of 0.5 mL/dose of Baiya SARS-CoV-2 Vax 2 (recombinant SARS-CoV-2 receptor-binding domain fused with FC region of human IgG1 vaccine)
  Arms: 50 μg Baiya SARS-CoV-2 Vax 2

SUMMARY:
The investigational product Baiya SARS-CoV-2 Vax 2 vaccine is a second-generation of protein subunit vaccine from plant. The primary objective aiming to evaluate the safety, tolerability, and reactogenicity of Baiya SARS-CoV-2 Vax 2 in adults (aged between 18 to 64 years, inclusive) after 2 doses of Baiya SARS-CoV-2 Vax 2 given 21 days apart IM, up to 28 days after the second vaccination. The secondary objective aiming to evaluate long-term safety profile (up to 1 year) and evaluate immunogenicity after 2 doses of Baiya SARS-CoV-2 Vax 2 given 21 days apart.

DETAILED DESCRIPTION:
The Baiya SARS-CoV-2 Vax 2 investigational vaccine is developed by Baiya Phytopharm Co., Ltd. for the active immunisation of adults against SARS-CoV-2, which causes coronavirus disease 2019 (COVID-19). This first in human (FIH) study will be conducted in healthy participants. Screening for the study will occur within a 42-day window prior to study enrolment. All eligible, consenting participants will receive Baiya SARS-CoV-2 Vax 2 vaccine at the assigned dose by IM injection, according to a repeat vaccination schedule (to be given 21 days apart). The study is an open-label, dose escalation, FIH study conducted in healthy adults aged 18 to 64 years (inclusive).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy man or woman between 18 to 64 years old (inclusive).
2. Give informed consent prior to study enrolment and all study procedures.
3. Participant must be able to comply with study procedures and be available for all study visits.
4. Participants must be in general good health based on medical history and physical examination as determined by the investigator(s) at Screening.
5. Males must be surgically sterile (>30 days since vasectomy with no viable sperm), practice true abstinence, or, if engaged in sexual activities with a female with childbearing potential, use condoms from first vaccination until 60 days after the last vaccination.
6. Females of child-bearing potential must practice true abstinence, or, if engaged in sexual activities with a male, agree to use highly effective (failure rate of <1% per year when used consistently and correctly), double-barrier contraceptive measures throughout the study and intend to continue use of contraception methods for at least 60 days following the last vaccination.
7. Female participants of childbearing potential must not be pregnant or breastfeeding.
8. Body temperature measured at forehead using validated device must be less than 37.5ºC at Screening.
9. Pulse must be no greater than 100 beats per minute at Screening.
10. Systolic blood pressure (SBP) must be between 90 to 160 millimetres of mercury (mmHg), inclusive, at Screening.
11. Participants must agree to refrain from donating blood, plasma, ovules, or sperm during the whole study.
12. Participants must have haematology, clinical chemistry, coagulation, and urinalysis test results that are not deviating from the normal reference range by age and gender or considered "not clinically significant" per investigator decision based on safety at Screening.
13. Female participants of child-bearing potential must have negative serum pregnancy test by beta human chorionic gonadotropin [β-HCG] at Screening and a negative urine-based pregnancy test within 24 hours prior to each investigational vaccine administration.
14. Women of non-child-bearing potential must:

    1. be classified as being postmenopausal (defined as having a history of amenorrhea for at least one year), or
    2. where history of amenorrhea is less than one-year, female participants must have a FSH level > 40 milli-international units per millilitre (mIU/mL), or
    3. have a physical examination for evidence of being surgically sterile (hysterectomy, bilateral oophorectomy, or salpingectomy).
15. All volunteers will be screened for serum antibodies against SARS-CoV-2 as evidence of previous infection using Enzyme-Linked Immunosorbent Assay (ELISA) and must have a negative result.

Exclusion Criteria:

1. Presence of clinically significant medical history, unstable chronic or acute disease, or physical or laboratory findings that in the opinion of the investigator(s) may potentially increase the expected risk of exposure to the investigational vaccine, compromise the safety of the participant, or interfere with any aspect of study conduct or interpretation of results. This will include any thrombocytopenia or bleeding disorder contraindicating IM vaccination.
2. Presence of self-reported or medically documented significant medical or psychiatric condition(s) as judged by the investigator(s) that it may not be in the participants' interest to participate in the study.
3. Presence of birthmarks, tattoos, wound, or other skin conditions over the deltoid region of both arms that in the opinion of the investigator, could reasonably obscure and interfere with evaluation of local ISRs.
4. Inadequate venous access to allow collection of blood samples.
5. Breastfeeding or planning to breastfeed from the time of the first vaccination to after the last vaccination, or pregnant as confirmed by a positive serum β-HCG pregnancy test at Screening or positive urine pregnancy test at subsequent clinic visits at timepoints as delineated in the schedule of assessments.
6. Received any prophylactic or therapeutic vaccine, or licensed or unlicensed vaccine, device, or blood product, within 4 weeks of first vaccination or 5 half-lives (whichever is longer) or anticipate doing so in the follow-up period defined for this study.
7. History of severe allergy (requiring hospital care), anaphylaxis, severe reaction to any drug or prior vaccination, or any known or suspected allergies or sensitivities to any component of the investigational vaccine or tobacco.
8. Participant is immunosuppressed as caused by disease (such as HIV)
9. Chronic use (more than 14 continuous days) of, or anticipated need to use, within the next 6 months of any medications that may be associated with impaired immune responsiveness or with immunosuppression.
10. History of hepatitis B or hepatitis C infection.
11. Receipt of immunoglobulins or blood products within 90 days of the first vaccination.
12. Receipt of other investigational products (drug, biologic, or device) within 60 days before the first vaccination.
13. History of alcohol or drug abuse that, in the opinion of the PI, could affect the participant's safety or compliance with study.
14. Participant is unwilling to abstain from blood donation during the course of the study, and/or is participating in any research study involving more blood sampling.
15. Participant is unwilling to abstain from donating plasma, ovules, sperm, or organs during the study.
16. Close contact with anyone known to have SARS-CoV-2 infection within 30 days prior to vaccine administration.
17. History of COVID-19 diagnosis.
18. On current treatment with investigational agents for prophylaxis of COVID-19 including COVID-19 Vaccine under EUA.
19. Planning to travel out of the country from enrolment through 29 days after the second vaccination.
20. Residing in a nursing home or other skilled nursing facility or having a requirement for skilled nursing care.
21. Is a participant at high risk of SARS-CoV-2 exposure in the opinion of the PI, including but not limited to an occupation (e.g., healthcare workers, active health care workers with direct patient contact, emergency response personnel) or close contact with a SARS-CoV-2 positive confirmed case (e.g., family member, housemate).
22. Presence of an acute illness, as determined by the participating Study Site investigator(s), with or without fever (forehead temperature measured with validated device ≥ 37.5 ºC) within 72 hours prior to each vaccination
23. Requirement for antipyretic or analgesic medication on a daily or every other day basis from enrolment through 72 hours after vaccination.
24. Current use of any prescription or over-the-counter medications within 7 days prior to vaccination, unless approved by the PI.
25. Has a positive result on SARS-CoV-2 antibody IgG/IgM measured by enzyme-linked immunosorbent assay (ELISA) at Screening.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-05-29 (Estimated); Study Completion 2024-04-10 (Estimated)

PRIMARY OUTCOMES:
Frequency and grade of solicited local and systemic reactogenicity AEs | 7-day post each vaccination
Frequency and grade of AEs | Post-vaccination - 28 days after second vaccination
Incidence of Serious Adverse Events (SAEs), Medically-Attended Adverse Events (MAAEs), and New-Onset Chronic Medical Conditions (NOCMCs) | Post-vaccination - 28 days after second vaccination
Changes in Blood Pressure (Systolic and Diastolic Blood Pressure) from Baseline | Post-vaccination - 28 days after second vaccination
  Blood pressure is measured mmHg. Blood pressure, both systolic and diastolic, at multiple timepoints according to the protocol will be compared to baseline value. Changes in blood pressure will be described using descriptive statistic (mean, standard deviation).
Changes in Pulse Rate from Baseline | Post-vaccination - 28 days after second vaccination
  Pulse rate is measured as beats per minute. Pulse rate at multiple timepoints according to the protocol will be compared to baseline value. Changes in pulse rate will be described using descriptive statistic (mean, standard deviation).
Changes in Respiratory Rate from Baseline | Post-vaccination - 28 days after second vaccination
  Respiratory rate is measured as breaths per minute. Respiratory rate at multiple timepoints according to the protocol will be compared to baseline value. Changes in respiratory rate will be described using descriptive statistic (mean, standard deviation).
Changes in Body Temperature from Baseline | Post-vaccination - 28 days after second vaccination
  Body temperature is measured as degree Celsius. Body temperature at multiple timepoints according to the protocol will be compared to baseline value. Changes in body temperature will be described using descriptive statistic (mean, standard deviation)
Changes in Physical Examinations from Baseline | Post-vaccination - 28 days after second vaccination
  Baseline physical examination will include head, ears, nose, throat, lungs, lymph nodes, heart, abdomen and skin. Symptom directed physical examination will be performed for each subsequent visit. Changes in physical conditions from baseline physical examination will be described.
Clinically relevant changes in haematology laboratory measurements | Up to 28 days after second vaccination
  Haematology laboratory value by Common Terminology Criteria for Adverse Event (CTCAE) scale version 5.0 (absolute and change from baseline where identified). The scale ranges from Grade 1 (Mild) to Grade 5 (Most Severe).
Clinically relevant changes in blood chemistry laboratory measurements | Up to 28 days after second vaccination
  Blood Chemistry laboratory value by Common Terminology Criteria for Adverse Event (CTCAE) scale version 5.0 (absolute and change from baseline where identified). The scale ranges from Grade 1 (Mild) to Grade 5 (Most Severe).
Clinically relevant changes in coagulation laboratory measurements | Up to 28 days after second vaccination
  Coagulation laboratory value by Common Terminology Criteria for Adverse Event (CTCAE) scale version 5.0 (absolute and change from baseline where identified). The scale ranges from Grade 1 (Mild) to Grade 5 (Most Severe).
Clinically relevant changes in urinalysis laboratory measurements | Up to 28 days after second vaccination
  Urinalysis laboratory value by Common Terminology Criteria for Adverse Event (CTCAE) scale version 5.0 (absolute and change from baseline where identified). The scale ranges from Grade 1 (Mild) to Grade 5 (Most Severe).
Treatment-emergent, clinically significant changes in Blood Pressure | Post-vaccination - 28 days after second vaccination
  Grade of treatment-emergent changes in blood pressure by Common Terminology Criteria for Adverse Event (CTCAE) scale version 5.0. The scale ranges from Grade 1 (Mild) to Grade 5 (Most Severe).
Treatment-emergent, clinically significant changes in Pulse Rate | Post-vaccination - 28 days after second vaccination
  Grade of treatment-emergent changes in pulse rate by Common Terminology Criteria for Adverse Event (CTCAE) scale version 5.0. The scale ranges from Grade 1 (Mild) to Grade 5 (Most Severe).
Treatment-emergent, clinically significant changes in Respiratory Rate | Post-vaccination - 28 days after second vaccination
  Grade of treatment-emergent changes in respiratory rate by Common Terminology Criteria for Adverse Event (CTCAE) scale version 5.0. The scale ranges from Grade 1 (Mild) to Grade 5 (Most Severe).
Treatment-emergent, clinically significant changes in Body Temperature | Post-vaccination - 28 days after second vaccination
  Grade of treatment-emergent changes in body temperature by Common Terminology Criteria for Adverse Event (CTCAE) scale version 5.0. The scale ranges from Grade 1 (Mild) to Grade 5 (Most Severe).
Treatment-emergent, clinically significant changes in Physical examinations | Post-vaccination - 28 days after second vaccination
  Baseline physical examination will include head, ears, nose, throat, lungs, lymph nodes, heart, abdomen and skin. Symptom directed physical examination will be performed for each subsequent visit. Grade of treatment-emergent changes by Common Terminology Criteria for Adverse Event (CTCAE) scale version 5.0. The scale ranges from Grade 1 (Mild) to Grade 5 (Most Severe).

SECONDARY OUTCOMES:
Frequency and Grade of Medically-Attended Adverse Events (MAAEs) | 28 days - 1 year after second vaccination
Frequency and Grade of New-Onset Chronic Medical Conditions (NOCMCs) | 28 days - 1 year after second vaccination
Incidence of SAEs | 28 days - 1 year after second vaccination
Geometric Mean Titer (GMT) of SARS-CoV-2 Specific Serum Neutralising Antibody | on 7, 14 and 28 days after second vaccination
  SARS-CoV-2 Specific Serum Neutralising Antibody as measured by Micro-neutralization assay, expressed as GMTs for each cohort
Geometric Mean Fold Rise (GMFR) of SARS-CoV-2 Specific Serum Neutralising Antibody | on 7, 14 and 28 days after second vaccination
  SARS-CoV-2 Specific Serum Neutralising Antibody as measured by Micro-neutralization assay, expressed as GMFRs for each cohort
Seroconversion Rate of SARS-CoV-2 Specific Serum Neutralising Antibody | on 7, 14 and 28 days after second vaccination
  Seroconversion Rate is defined as the proportion of participants who achieves a greater than or equal to 4-fold rise in SARS-CoV-2 specific serum neutralising antibody level from baseline
Geometric Mean Titer (GMT) of SARS-CoV-2 Surrogate Viral Neutralising Antibody | on 7, 14 and 28 days after second vaccination
Geometric Mean Fold Rise (GMFR) of SARS-CoV-2 Surrogate Viral Neutralising Antibody | on 7, 14 and 28 days after second vaccination
Seroconversion Rate of SARS-CoV-2 Surrogate Viral Neutralising Antibody | on 7, 14 and 28 days after second vaccination
  Seroconversion Rate is defined as a greater than or equal to 4-fold rise in SARS-CoV-2 surrogate viral neutralising antibody from baseline
Geometric Mean Titer (GMT) of RBD-specific IgG Antibody | on 7, 14 and 28 days after second vaccination
  Measured by enzyme-linked immunosorbent assay (ELISA)
Geometric Mean Fold Rise (GMFR) of RBD-specific IgG Antibody | on 7, 14 and 28 days after second vaccination
  Measured by enzyme-linked immunosorbent assay (ELISA)
Seroconversion Rate of RBD-specific IgG Antibody | on 7, 14 and 28 days after second vaccination
  Measured by enzyme-linked immunosorbent assay (ELISA). Seroconversion Rate is defined as a greater than or equal to 4-fold rise in RBD-specific IgG Antibody from baseline
Percentage of participants who have positive RBD-specific CD4+ and CD8+ T-cell IFN-y ELISpot responses | on 7, 14 and 28 days after second vaccination
  Measured by IFN-y ELISpot assay
Median number of spot-forming cells (SFC) per 1 million PBMCs | on 7, 14 and 28 days after second vaccination
  Measured by IFN-y ELISpot assay
Percentage of participants who shows positive specific T-helper 1 responses, or T-helper 2 responses | on 7, 14 and 28 days after second vaccination
  Quantified by Intracellular Cytokine Staining
Median percentage of specific T-helper 1 responses and T-helper 2 responses ratio | on 7, 14 and 28 days after second vaccination
  Quantified by Intracellular Cytokine Staining

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Saovabha Memorial Institute, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No